CLINICAL TRIAL: NCT00889291
Title: HeRO Vascular Access Device Post Market Procedural Survey Protocol
Acronym: PPS
Status: Completed | Type: Observational
Sponsor: Merit Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 1-Abbs
Record Dates: First submitted 2009-04-09; First posted 2009-04-28 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: End Stage Renal Disease
Keywords: End stage renal disease; Bacteremia; HeRO Vascular Access Device; Access challenged; Catheter dependent; End stage renal disease requiring vascular access. See HeRO device instructions for use for appropriate patient population
MeSH Terms: conditions — Kidney Failure, Chronic; Bacteremia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
Post market observational survey of a vascular access device for access-challenged patients. Data collection efforts focused on patient medical and access history and implant procedure results.

DETAILED DESCRIPTION:
Evaluation Design: This is a multi-center post market observational survey designed to collect procedural data on a minimum of 50 HeRO™ patients in the commercialization phase. Data will be collected retrospectively for patients already implanted with the HeRO™ device in the commercialization phase or prospectively for patients that receive the HeRO™ Device during the data collection period. No special patient screening, testing, or procedures are required. There is no required patient follow-up.

Subject Population: Any patients the investigator deems/deemed eligible for HeRO™ implant with complete procedural data are eligible for inclusion in this post market observational survey.

Endpoints: None

Inclusion/Exclusion Criteria: There are no formal screening criteria other than patients must have all required procedural data points available for recording on the case report form.

ELIGIBILITY:
Inclusion Criteria:

* None

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: End stage renal disease patients requiring vascular access
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2008-12; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Device placement success | End of procedure

CONTACTS AND LOCATIONS:
Overall Officials: Marc Glickman, MD, Principal Investigator — Sentara Heart Hospital, Norfolk, VA

REFERENCES:
- See also: Additional information regarding the HeRO Vascular Access Device — http://www.hemosphere.net/